CLINICAL TRIAL: NCT04617470
Title: Niraparib as Maintenance Treatment in Platinum Responsive Ovarian Cancer Patients: a Real Life Study by MITO Group
Brief Title: Niraparib as Maintenance Treatment in Platinum Responsive Ovarian Cancer Patients: a Real Life Study
Acronym: MITO 34
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 2487
Record Dates: First submitted 2020-10-05; First posted 2020-11-05 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational phase IV study evaluating Niraparib as maintenance treatment in patients with platinum sensitive, platinum responsive, recurrent ovarian cancer in a real life setting.

DETAILED DESCRIPTION:
This is an observational phase IV study evaluating Niraparib as maintenance treatment in patients with platinum sensitive, platinum responsive, recurrent ovarian cancer in a real life setting. Will be enrolled all patients who have been part of the Italian Compassionate Use Program (CUP) prior to participating in this study. Once the CUP will be closed the trial will continue with th prospective collection of data of patients treated with Niraparib according to the label for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* patients that received niraparib as monotherapy for the maintenance treatment of platinum-sensitive, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer after response (complete or partial) to platinum-based chemotherapy as part of the CUP, regardless of whether the patient is receiving niraparib at the time of enrolment;
* patients with high grade serous ovarian cancer treated with Niraparib according to the label will be included;
* patients able to understand the study procedures and that agree to participate in the study by providing written informed consent

Exclusion Criteria:

No exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with platinum-sensitive, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to two years
  To compare PFS of patients with advanced, platinum sensitive ovarian cancer treated with Niraparib as maintenance treatment

SECONDARY OUTCOMES:
TFST | up to two years
  Time to first subsequent therapy
TSST | up to two years
  Time to second subsequent therapy
OS | up to two years
  Overall Survival
ORR | up to two years
  Overall Response Rate
Incidence of treatment-emergent adverse events | up to two years
  Toxicity will be evaluated by NCI CTCAE V 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy